CLINICAL TRIAL: NCT00071903
Title: The Role of Susceptibility to Thrombosis in the Pseudotumor Cerebri of Nephropathic Cystinosis: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040010; 04-CH-0010
Record Dates: First submitted 2003-11-03; First posted 2003-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-18

CONDITIONS: Pseudotumor Cerebri; Cystinosis
Keywords: Thrombophilia; Idiopathic Intracranial Hypertension; Kidney Involvement; Lysosomal Storage Disorder; Cystine; Pseudotumor Cerebri; Susceptibility to Thrombosis; Nephropathic Cystinosis; PTC; Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri; Cystinosis; Thrombophilia; Lysosomal Storage Diseases; Intracranial Hypertension

SUMMARY:
This study will examine whether the tendency to have thrombosis, or the formation of blood clots inside blood vessels, has a role in the development of pseudotumor cerebri (PTC). PTC causes symptoms and signs of isolated elevated blood pressure in the cranium, or covering of the brain. The disorder can lead to significant, negative effects on the visual system. Increased pressure of the cerebrospinal fluid, that is, fluid around the brain, is a factor, but the cause of the disorder is not clear. There has been documentation of clustering of PTC within families. It suggests that potential genetic polymorphisms-abilities to take on different forms-may become evident after exposure to conditions known to trigger PTC.

Thrombosis comes about by interactions between genetic and environmental or acquired factors, or both, resulting in a blood clot at a specific time and location. Because the disease occurs in episodes, the interaction of the genetic and nongenetic risk factors is important. Cystinosis is a recessive disorder caused by deposits of cystine within the lysosomes of cells-that is, sac-like cell parts that contain various enzymes. Involvement of the kidneys remains the primary characteristic, eventually leading to renal failure. Of all of the risk factors that make it easier for blood clotting, a high level of a substance called homocysteine is of particular interest. Too much homocysteine in blood plasma is a common finding in patients with kidney failure, and it has been recently identified as an independent risk factor for diseases of the blood vessels.

Participants of all ages who meet the Dandy criteria for PTC may be eligible for this study. Pregnant women will be excluded. There will also be a control group of nephropathic cystinosis patients who do not have PTC.

Participants will be asked to undergo the following tests and procedures:

* Medical history.
* Physical examination, to evaluate the eye and nervous systems.
* Collection of blood for DNA and other tests.
* Collection of cerebrospinal fluid, through a procedure called lumbar puncture or spinal tap.

The evaluation of patients will generally last 3 to 4 days. For the collection of cerebrospinal fluid, the patient's skin on the back will be numbed with a local anesthetic. A special needle will be inserted into the back, and a small amount of the fluid will be drawn through the needle. There will be pain for a minute, although there can be a headache lasting 24 hours. Also, there may be bruising, local pain, bleeding, or infection where the needle enters. Patients may also have a magnetic resonance imaging scan of their head. During the MRI scan, patients will lie still on a table that slides in and out of a metal cylinder surrounded by a strong magnetic field. Patients will be able to communicate with the MRI staff at all times and may ask to be moved out of the machine at any time.

DETAILED DESCRIPTION:
During the follow-up of cystinosis patients under protocol #78-HG-0093 "Use of Cysteamine in the Treatment of Cystinosis", we found that 6 of our NIH patients developed papilledema and were diagnosed with pseudotumor cerebri (PTC), whose occurrence has not been previously reported in cystinosis. The goal of this protocol is to identify the role of thrombosis susceptibility in the development of PTC in nephropathic cystinosis patients in view of our recent findings regarding genetic susceptibility to thrombosis in PTC in general. We propose a case-control study. A total of 9 nephropathic cystinosis patients who developed PTC and 9 control nephropathic cystinosis patients without PTC will be screened based upon a thrombosis susceptibility screening panel, including total homocysteine, protein C and S, antithrombin III, fibrinogen, Factor VIII, Factor IX, Factor XI levels, testing for PT, PTT, activated protein C resistance, antiphospholipid antibodies (ACA panel and Lupus AC) and screening for FV Leiden mutation, FV G1628A polymorphism, FV R2 allele, Prothrombin 20210 mutation and 5,10-methylenetetrahydrofolate reductase (MTHFR) gene C677T polymorphism in patients with severe homocysteinemia (greater than or equal to 100 micro mol/l).

We will compare the prevalence of the factors that lead to thrombosis susceptibility in the cases and controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

The inclusion criteria include only a confirmed diagnosis of pseudotumor cerebri (past or present) in a patient with nephropathic cystinosis. Patients will be diagnosed as having pseudotumor cerebri based upon modified Dandy criteria:

1. signs and symptoms related to increased intracranial pressure;
2. no localizing neurological signs with the exception of unilateral or bilateral sixth nerve palsy;
3. neuroimaging study showing no mass lesion or hydrocephalus;
4. elevated opening pressure with normal cerebrospinal fluid contents on lumbar puncture.

Nephropathic cystinosis patients of all ages who meet the Dandy criteria for PTC will be considered for the study.

EXCLUSION CRITERIA:

Pregnant patients will be excluded from the study.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18
Dates: Start 2003-10-30; Study Completion 2008-07-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Quattrone A, Gambardella A, Carbone AM, Oliveri RL, Lavano A, De Marco EV, Civitelli D, Bono F, Zappia M, Pardatscher K, DiMinno G. A hypofibrinolytic state in overweight patients with cerebral venous thrombosis and isolated intracranial hypertension. J Neurol. 1999 Nov;246(11):1086-9. doi: 10.1007/s004150050517. PMID 10631643
- [Background] Martins AN. Resistance to drainage of cerebrospinal fluid: clinical measurement and significance. J Neurol Neurosurg Psychiatry. 1973 Apr;36(2):313-8. doi: 10.1136/jnnp.36.2.313. PMID 4541080
- [Background] Calabrese VP, Selhorst JB, Harbison JW. CSF infusion test in pseudotumor cerebri. Trans Am Neurol Assoc. 1978;103:146-50. No abstract available. PMID 757043